CLINICAL TRIAL: NCT03335046
Title: Project HOMES: Home Visits to Optimize Medical and Educational Success
Brief Title: Home Visits to Optimize Medical and Educational Success Among Sacramento Schoolchildren With Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1114637
Record Dates: First submitted 2017-11-03; First posted 2017-11-07 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Asthma; Chronic School Absenteeism
Keywords: Home Visit; School Absenteeism
MeSH Terms: conditions — Asthma | interventions — House Calls; Standard of Care

STUDY DESIGN:
Intervention Model Description: The study will be a randomized wait-list control trial. Participants will be randomized to the intervention or control arm for the study observation period. At the conclusion of the observation period, the control group will receive the intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention arm will receive the home visit intervention, consisting of 2 visits to the home by a team consisting of a pediatric medical provider and a school teacher or school support staff member. This team will evaluate the child's home environment to assess for potential asthma triggers that may lead to school absenteeism, and provide strategies and material goods to help reduce those triggers.
  Interventions: Behavioral: Home Visit
- Wait-List Control (Other): The control group will receive standard interventions carried out by the school system for students at risk for chronic absenteeism. Following the study observation period, this control group will then receive the home visits performed for the intervention group.
  Interventions: Behavioral: Home Visit; Behavioral: Standard Care

INTERVENTIONS:
Behavioral: Home Visit — The intervention will consist of a series of home visitations to chronically absent students with co-morbid asthma. These visits will consist of a home environment evaluation, medication adherence and knowledge assessment, distribution of home environmental allergen reduction items such as mattress and pillow encasements, as well as review and reinforcement of any asthma action plans or care plans provided by patient's primary care physicians or medical home.
Behavioral: Standard Care — Standard care will refer to the procedures carried out by the school district to address students with chronic absenteeism. This includes parent-teacher and parent-school administrator meetings and communications and may also include home visits carried out by classroom teachers or student support center staff.
  Arms: Wait-List Control

SUMMARY:
This study will establish a multi-disciplinary home visitation team consisting of a medical provider and school teacher or staff member, and will evaluate whether a series of visits from this team will help decrease school absenteeism among children with asthma.

ELIGIBILITY:
Inclusion Criteria:

* Students in elementary school (K-6) in the Sacramento City Unified School District
* Identified as at risk for chronic absenteeism based on previous year and/or first 8 weeks of school year
* Have a current diagnosis of asthma

Exclusion Criteria:

* Underlying chronic conditions such as cystic fibrosis, chronic lung disease with oxygen dependence, immunodeficiency syndromes

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Missed School Days | One academic year
  The number of school days missed over the course of an academic year

SECONDARY OUTCOMES:
Healthcare Utilization | One academic year
  Number of emergency department or urgent care visits for asthma
Asthma Symptom Report | One academic year
  Patient and family self-report of number of days where asthma symptoms were experienced, collected monthly
Asthma Control Test | One academic year
  Numeric score from the Childhood Asthma Control Test, collected monthly

CONTACTS AND LOCATIONS:
Locations (1):
- University of California Davis, Sacramento, California, United States